CLINICAL TRIAL: NCT01764022
Title: Multicenter Randomized Double-blind Phase III Clinical Trial Comparing Safety and Efficacy of BCD-022 (CJSC BIOCAD, Russia) Used With Paclitaxel to Herceptin® Used With Paclitaxel in the First-line Treatment of HER2+ Metastatic Breast Cancer Patients
Brief Title: A Safety and Efficacy Study of BCD-022 With Paclitaxel Compared to Herceptin With Paclitaxel in HER2+ Metastatic Breast Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCD-022-02
Record Dates: First submitted 2013-01-07; First posted 2013-01-09 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Human Epithelial Receptor (HER)-2 Positive Breast Cancer
Keywords: breast cancer; trastuzumab
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BCD-022 (Experimental): BCD-022 is a product code for trastuzumab biosimilar manufactured by CJSC BIOCAD, Russia. In this arm patients will receive 6 courses of treatment with BCD-022 in combination with paclitaxel. Patients will receive BCD-022 at a loading dose of 8 mg/kg (once), followed by maintenance dose of 6 mg/kg every 3 weeks (5 administrations), + paclitaxel 175 mg/m2 every 3 weeks as 3 hour intravenous infusion (6 administrations).
  Interventions: Drug: Trastuzumab; Drug: Paclitaxel
- Herceptin® (Active Comparator): In this arm patients will receive 6 courses of treatment with Herceptin® (F. Hoffmann-La Roche Ltd., Switzerland) in combination with paclitaxel. Patients will receive Herceptin® at a loading dose of 8 mg/kg (once), followed by maintenance dose of 6 mg/kg every 3 weeks (5 administrations), + paclitaxel 175 mg/m2 every 3 weeks as 3 hour intravenous infusion (6 administrations).
  Interventions: Drug: Trastuzumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Trastuzumab — Patients will receive 6 courses of trastuzumab in combination with paclitaxel. Trastuzumab will be administered at a loading dose of 8 mg/kg (once), followed by maintenance dose of 6 mg/kg every 3 weeks (5 administrations) as 90 min intravenous infusion every 3 weeks (on Day 1 of each cycle).
  Other Names: BCD-022; Herceptin
Drug: Paclitaxel — Paclitaxel will be administered at a dose of 175 mg/m2 every 3 weeks (on Day 1 of each course) as 3 hour intravenous infusion (6 courses totally).
  Other Names: Taxacad

SUMMARY:
BCD-022-02 is a double-blind randomized clinical trial comparing efficacy of BCD-022 (INN: trastuzumab) and paclitaxel to Herceptin and paclitaxel in HER2-positive metastatic breast cancer with pharmacokinetics substudy. The purpose of the study is to demonstrate the non-inferiority of efficacy and safety of BCD-022 compared to Herceptin. Also study includes pharmacokinetics assessment.

DETAILED DESCRIPTION:
The study is based on the hypothesis of equivalence of BCD-022 (trastuzumab by JSC BIOCAD, Russia) in combination with paclitaxel used as the therapy of inoperable or metastatic HER2(+) breast cancer in comparison with Herceptin® (F. Hoffmann-La Roche Ltd., Switzerland) in combination with paclitaxel. The objectives of the study is to evaluate efficacy, safety and pharmacokinetics of BCD-022 compared with reference trastuzumab by 1. overall response rate and other efficacy parameters; 2. incidence and severity of adverse events; 3. serum concentration after the first and multiple trastuzumab administration; 4. incidence and concentration of anti-trastuzumab antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and ability to follow the Protocol procedures;
* Age from 18 years to 75 years inclusive;
* Female gender;
* Histologically confirmed breast cancer (BC);
* Metastatic BC (stage IV according to TNM classification version 6);
* Grade 3+ HER2 overexpression confirmed by immunohistochemical (IHC) staining or grade 2+ HER2 overexpression accompanied by HER2 gene amplification confirmed by fluorescent hybridization in situ (FISH) ;
* Documented results of oestrogen and progesterone receptors expression analysis;
* Eastern Cooperative Oncology Group (ECOG) status 0, 1 or 2, not increasing within 2 weeks prior to randomization;
* Life expectancy - 20 weeks or more from the moment of randomization;
* Presence of at least 1 tumour with a size not less than 1 cm (revealed with computed tomography (CT) slice thickness not more than 5 mm). Patients having bone metastasis as the only measurable tumour are not eligible for the trial;
* Patients of childbearing potential must implement reliable contraceptive measures during the study treatment, starting 4 weeks prior to inclusion into the trial and until 6 months after the last administration of the study drug.

Exclusion Criteria:

* Previous anticancer therapy for metastatic BC, including cytotoxic chemotherapy, or previous anticancer therapy with signal transduction inhibitors (e.g. lapatinib), biological drugs (e.g. trastuzumab, bevacizumab), experimental (not approved for BC therapy) anticancer drugs. Any previous hormonal therapy is allowed;
* Disease progression within 6 months after adjuvant and/or neoadjuvant anti BC therapy;
* Surgery, radiation therapy, use of any experimental medications within 4 weeks (28 days) prior to randomization;
* Hypersensitivity to paclitaxel and all medications containing polyoxyethylated castor oil, hypersensitivity to dexamethasone, diphenhydramine, ranitidine/cimetidine, recombinant murine proteins, contrast agents or excipients of study medications;
* BC metastases in central nervous system, progressing or clinically manifested (e.g. cerebral oedema, spinal cord injury), with exception of non-progressing metastases not requiring treatment with glucocorticosteroids and/or anticonvulsants within 4 weeks prior to randomization;
* Cardiovascular system pathology (congestive heart failure (CHF) stage III-IV according to New York Heart Association (NYHA) classification, unstable angina pectoris, myocardial infarction) within 12 months prior to randomization;
* Uncontrolled hypertension comprising all cases of arterial hypertension when no decrease in blood pressure could be achieved despite treatment with a combination of 3 antihypertensive drugs including one diuretic and non-medicamental correction methods (low salt diet, physical exercise);
* Left ventricular ejection fraction <50% according to electrocardiography;
* Neutrophils ≤1500/mm3;
* Platelets ≤100 000/mm3;
* Hemoglobin ≤90 g/L;
* Creatinine level ≥ 1.5 × upper limit of normal (ULN);
* Bilirubin level ≥ 1.5 × ULN;
* Asparagine transferase (AST) and alanine transferase (ALT) levels ≥ 2.5 × ULN (5 × ULN for patients with liver metastases);
* Alkaline phosphatase level ≥ 5 × ULN;
* Pregnancy or lactation;
* Any other concomitant cancer including contralateral breast cancer revealed within 5 years prior to screening, except curatively treated intraductal carcinoma in situ, curatively treated cervical carcinoma in situ or curatively treated basal cell or squamous cell carcinoma;
* Conditions limiting patient's adherence to protocol requirements (dementia, neurologic or psychiatric disorders, drug addiction, alcoholism and others);
* Stage II-IV neuropathy according to Common Terminology Criteria for Adverse Events (CTCAE) v.4.0;
* Concomitant participation in other clinical trials, previous participation in other clinical trials within 30 days before entering into the trial, previous participation in the same trial;
* Acute or active chronic infections;
* Hepatitis C virus, hepatitis B virus, HIV or syphilis infections;
* Obstacles in intravenous administration of study drugs

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2012-10; Primary Completion 2015-03 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ivanov, MD, PhD, Study Chair — Vice-president, R&D
Locations (36):
- Belarus (4):
  - Brest Region Clinical Oncology Dispensary, Brest
  - Grodno Regional Hospital, Grodno
  - Gomel Region Clinical Oncology Dispensary, Homyel
  - Vitebsk State Medical University of Order of Peoples' Friendship, Vitebsk
- India (3):
  - HCG Bangalore Institute of Oncology, Bangalore
  - M.S.Ramaiah Memorial Hospital, Bangalore
  - Narayana Hrudayalaya Hospitals, Bangalore
- Russia (20):
  - State Health Institution of Moscow "Moscow City Oncology Hospital #62 of Moscow Board of Health", Stepanovskoye, Moscow Oblast
  - Arkhangelsk District Clinical Oncology Dispensary, Arkhangelsk
  - Non-governmental Healthcare Institution "Railway Clinical hospital on the Chelyabinsk Station of JSC Russian Railways", Chelyabinsk
  - State-financed Health Institution "Chelyabinsk Region Clinical Oncology Dispansary", Chelyabinsk
  - State-financed Health Institution "Republican Clinical Oncology Hospital", Izhevsk
  - Institution of Russian Academy of Medical Sciences "Russian Cancer Research Center named after N.N. Blokhin", Moscow
  - Federal State Institution "Moscow Institute of Cancer Research named after P.A. Hertsen" Ministry of Health of Russian Federation, Moscow
  - Regional State Health Institution "Orlov Oncology Dispansary", Oryol
  - State Health Institution "Region Oncology Dispansary", Penza
  - Perm Region Oncology Dispensary, Perm
  - Federal Government Budgetary Institution "Rostov Institute of Cancer Research" of Ministry of Health of Russian Federation, Rostov-on-Don
  - Military Medical Academy named after S.M. Kirov, Saint Petersburg
  - Saint Petersburg City Clinical Oncology Center, Saint Petersburg
  - N.N.Petrov Oncology Research Center, Saint Petersburg
  - Russian scientific center of radiology and surgery technologies, Saint Petersburg
  - State-financed Health Institution "Samara Region Clinical Oncology Dispansary", Samara
  - Oncology Dispensary 2, Sochi
  - State-financed Health Institution "Stavropol Region Clinical Oncology Dispansary", Stavropol
  - Republican Clinical Oncology Dispensary of Ministry of Health republic Bashkortostan, Ufa
  - Volgograd District Oncology Dispensary №1, Volgograd
- Ukraine (9):
  - Donetsk City Oncology Dispensary, Donetsk
  - Donetsk Regional Antitumor Center, Donetsk
  - Kharkiv Regional Clinical Oncology Center, Kharkiv
  - Kryvyi Rih Oncology Dispensary, Kryvyi Rih
  - Lviv Regional State Cancer Diagnostics and Treatment Center, Lviv
  - City Hospital №2, Makiivka
  - Poltava Regional Clinical Oncology Dispensary, Poltava
  - Zakarpatskyi Regional Clinical Oncology Center, Uzhhorod
  - Vinnytsia Regional Clinical Oncology Dispensary, Vinnytsia

REFERENCES:
- [Derived] Alexeev SM, Khorinko AV, Mukhametshina GZ, Shelepen KG, Burdaeva ON, Kulik SA, Satheesh CT, Srivastava K, Vikranth M, Kryukov F, Paltusova AN, Shustova MS, Ivanov RA. Randomized double-blind clinical trial comparing safety and efficacy of the biosimilar BCD-022 with reference trastuzumab. BMC Cancer. 2020 Aug 20;20(1):783. doi: 10.1186/s12885-020-07247-9. PMID 32819305

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In BCD-022 group 2 patients were exluded from any analysis due to:
  * Death prior to the first drug administration
  * Informed consent withdrawal prior to the first drug administration
Groups:
- BCD-022 (CJSC BIOCAD): BCD-022 is a product code for trastuzumab biosimilar manufactured by CJSC BIOCAD, Russia. In this arm patients will receive 6 courses of treatment with BCD-022 in combination with paclitaxel. Patients will receive BCD-022 at a loading dose of 8 mg/kg (once), followed by maintenance dose of 6 mg/kg every 3 weeks (5 administrations), + paclitaxel 175 mg/m2 every 3 weeks as 3 hour intravenous infusion (6 administrations).
- Herceptin ® (F. Hoffmann-La Roche Ltd., Switzerland): In this arm patients will receive 6 courses of treatment with Herceptin in combination with paclitaxel. Patients will receive Herceptin at a loading dose of 8 mg/kg (once), followed by maintenance dose of 6 mg/kg every 3 weeks (5 administrations), + paclitaxel 175 mg/m2 every 3 weeks as 3 hour intravenous infusion (6 administrations).
Period: Overall Study
Arm/Group | BCD-022 (CJSC BIOCAD) | Herceptin ® (F. Hoffmann-La Roche Ltd., Switzerland)
Started | 115 | 110
Received at Least 1 Dose of Study Drug | 113 | 110
Completed (Received 6 cycles of therapy during main period of the study or had disease progression) | 107 | 96
Not Completed | 8 | 14
Not completed — Death | 3 | 5
Not completed — Withdrawal by Subject | 2 | 6
Not completed — Lack of Efficacy | 0 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Population: 223 of 225 randomized patients received at least one BCD-022 or Herceptin® injection. 2 patients were excluded prior to first drug administration. Patients who do not received at least one study drug administration were not included to any analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | BCD-022 (CJSC BIOCAD) | Herceptin ® (F. Hoffmann-La Roche Ltd., Switzerland) | Total
Number analyzed (Participants) | 115 | 110 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.687 (10.948) | 50.573 (9.877) | 50.63 (10.415)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 110 | 225
  Male | 0 | 0 | 0
HER2 Expression [Count of Participants; unit: Participants]
  HER2 +++ | 100 | 97 | 197
  HER2 ++ | 14 | 13 | 27
  Unknown | 1 | 0 | 1
Histologic type of cancer [Count of Participants; unit: Participants]
  Ductal | 36 | 33 | 69
  Medullar | 3 | 4 | 7
  Lobular | 23 | 18 | 41
  Tubular | 35 | 37 | 72
  Mucinouse | 3 | 5 | 8
  Micropapillary | 1 | 0 | 1
  Unknown histilogic type | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
  The response was assessed at the screening, after 3 therapy cycles and after 6 therapy cycles. If CT after 3 or 6 therapy cycles revealed the complete or partial response, a confirmatory CT scan was performed 4 weeks later. The best response during the study was assessed.
Time Frame: Day 127
Population: The population for efficacy analysis included patients who received at least one injection of study drug and had evaluable results of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-022 (CJSC BIOCAD) | Herceptin ® (F. Hoffmann-La Roche Ltd., Switzerland)
Number analyzed (Participants) | 113 | 110
Participants | 56 | 48

2. Primary Outcome: Area Under the Curve After the First Test Drug Administration
Description: Primary outcome measure for pharmacokinetics (PK) substudy. AUC(0-504) of trastuzumab in HER2(+) mBC patients after first administration of BCD-022 with paclitaxel or Herceptin® with paclitaxel.
Time Frame: up to Day 22, after the first trastuzumab administration (time points for blood samples: 0 h 1.5 h, 3 h, 4.5 h, 6 h, 24 h, 96 h, 168 h, 336 h and 504 h)
Population: Patients who received one dose of study drug and after 504 hours after the injection had missed <= 1 blood sample collection to analyse pharmacokinetics.
Measure: Median (Inter-Quartile Range); unit: (ng/ml)*hour
Arm/Group | BCD-022 (CJSC BIOCAD) | Herceptin ® (F. Hoffmann-La Roche Ltd., Switzerland)
Number analyzed (Participants) | 107 | 104
(ng/ml)*hour | 28969372.5 [20165337.0 to 36096712.5] | 28796527.9 [20430685.5 to 36232918.5]

3. Secondary Outcome: Complete Response Rate
Description: as for outcome 1
Time Frame: Day 127
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-022 (CJSC BIOCAD) | Herceptin ® (F. Hoffmann-La Roche Ltd., Switzerland)
Number analyzed (Participants) | 113 | 110
Participants | 4 | 2

4. Secondary Outcome: Partial Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
  The response was assessed at the screening, after 3 therapy cycles and after 6 therapy cycles. If CT after 3 or 6 therapy cycles revealed the complete or partial response, a confirmatory CT scan was performed 4 weeks later. The best response during the study was assessed.
Time Frame: Day 127
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-022 (CJSC BIOCAD) | Herceptin ® (F. Hoffmann-La Roche Ltd., Switzerland)
Number analyzed (Participants) | 113 | 110
Participants | 52 | 46

5. Secondary Outcome: Stabilization Rate
Description: as for outcome 1
Time Frame: Day 127
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-022 (CJSC BIOCAD) | Herceptin ® (F. Hoffmann-La Roche Ltd., Switzerland)
Number analyzed (Participants) | 113 | 110
Participants | 28 | 21

6. Secondary Outcome: Progression Rate
Description: as for outcome 1
Time Frame: Day 127
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | BCD-022 (CJSC BIOCAD) | Herceptin ® (F. Hoffmann-La Roche Ltd., Switzerland)
Number analyzed (Participants) | 113 | 110
Participants | 25 | 28

7. Secondary Outcome: Treatment Postponed Due to AE/SAE
Description: Secondary outcome measure for safety evaluation
Time Frame: Day 127
Population: Patients who received at least one injection of study drug.
Measure: Number; unit: participants
Arm/Group | BCD-022 (CJSC BIOCAD) | Herceptin ® (F. Hoffmann-La Roche Ltd., Switzerland)
Number analyzed (Participants) | 113 | 110
participants | 4 | 5

8. Secondary Outcome: Treatment Discontinuation Due to AE/SAE
Description: Secondary outcome measure for safety evaluation
Time Frame: Day 127
Population: Patients who received at least one injection of study drug.
Measure: Number; unit: participants
Arm/Group | BCD-022 (CJSC BIOCAD) | Herceptin ® (F. Hoffmann-La Roche Ltd., Switzerland)
Number analyzed (Participants) | 113 | 110
participants | 0 | 1

9. Secondary Outcome: Occurrence of Neutralizing Anti-trastuzumab Antibodies
Description: Secondary outcome measure for immunogenicity assessment. Patient was suggested as NAB-positive if neutralizing anti-trastuzumab antibodies were detected at any of the specified timepoints. Total number of NAB-positive patients in each are presented.
Time Frame: Day 1 (before the drug administration), Day 14, 64, 127 and 154
Population: Patients who received at least one injection of study drug
Measure: Number; unit: participants
Arm/Group | BCD-022 (CJSC BIOCAD) | Herceptin ® (F. Hoffmann-La Roche Ltd., Switzerland)
Number analyzed (Participants) | 113 | 110
participants | 3 | 4

10. Secondary Outcome: Cmax After the First Test Drug Administration
Description: Secondary outcome measure for PK substudy. Peak serum concentration of trastuzumab after single administration of BCD-022 + paclitaxel or Herceptin® + paclitaxel
Time Frame: Up to Day 22
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | BCD-022 (CJSC BIOCAD) | Herceptin ® (F. Hoffmann-La Roche Ltd., Switzerland)
Number analyzed (Participants) | 107 | 104
ng/ml | 218720.0 [178270.0 to 264700.0] | 216710.0 [186740.0 to 269780.0]

11. Secondary Outcome: Tmax After the First Test Drug Administration
Description: Secondary outcome measure for PK substudy. Time to reach peak serum concentration of trastuzumab after the first administration of BCD-022 + paclitaxel or Herceptin® + paclitaxel
Time Frame: Up to Day 22
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | BCD-022 (CJSC BIOCAD) | Herceptin ® (F. Hoffmann-La Roche Ltd., Switzerland)
Number analyzed (Participants) | 107 | 104
hours | 160.6 [103.2 to 207.6] | 162.1 [101.9 to 201.6]

12. Secondary Outcome: T1/2 After the First Test Drug Administration
Description: Secondary outcome measure for PK substudy. Half-life period of trastuzumab after the first administration of BCD-022 + paclitaxel or Herceptin® + paclitaxel.
Time Frame: Up to Day 22
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Herceptin ® (F. Hoffmann-La Roche Ltd., Switzerland) | BCD-022 (CJSC BIOCAD)
Number analyzed (Participants) | 104 | 107
hours | 162.1 [101.9 to 201.6] | 160.6 [103.2 to 207.6]

13. Secondary Outcome: Cmax After the Sixth Test Drug Administration
Description: Secondary outcome measure for PK substudy. Peak serum concentration of trastuzumab after the sixth administration of BCD-022 + paclitaxel or Herceptin® + paclitaxel.
Time Frame: Up to Day 127
Population: Patients who received six dose of study drug and had missed <= 1 blood sample collection to analyse pharmacokinetics.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | BCD-022 (CJSC BIOCAD) | Herceptin ® (F. Hoffmann-La Roche Ltd., Switzerland)
Number analyzed (Participants) | 36 | 33
ng/ml | 168735.0 [148810.0 to 204870.0] | 169220.0 [150140.0 to 179230.0]

14. Secondary Outcome: Tmax After the Sixth Test Drug Administration
Description: Secondary outcome measure for PK substudy. Time to reach peak serum concentration of trastuzumab after the sixth administration of BCD-022 + paclitaxel or Herceptin® + paclitaxel
Time Frame: Up to Day 127
Population: Patients who received six dose of study drug and had missed <= 1 blood sample collection to analyse pharmacokinetics.
Measure: Median (Inter-Quartile Range); unit: hour
Arm/Group | BCD-022 (CJSC BIOCAD) | Herceptin ® (F. Hoffmann-La Roche Ltd., Switzerland)
Number analyzed (Participants) | 36 | 33
hour | 185.8 [146.3 to 237.1] | 192.9 [137.9 to 237.1]

ADVERSE EVENTS:
Time Frame: up to 154 days
Description: Population for safety analysis included patients who received at least one injection of study drug (n=223).
Arm/Group | BCD-022 (CJSC BIOCAD) | Herceptin ® (F. Hoffmann-La Roche Ltd., Switzerland)
All-Cause Mortality (participants affected / at risk) | 3/113 | 5/110
Serious Adverse Events (participants affected / at risk) | 8/113 | 13/110
Other Adverse Events (participants affected / at risk) | 106/113 | 104/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BCD-022 (CJSC BIOCAD) (N=113) | Herceptin ® (F. Hoffmann-La Roche Ltd., Switzerland) (N=110)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 — lethal outcome
Death for unknown reason (General disorders) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 — lethal outcome
Paroxism of atrial fibrillation (Cardiac disorders) | 0 | 2
Ventricular extrasystolone RYAN-1 (Cardiac disorders) | 0 | 1
Anemia with trombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Diarrhea with vomiting and weakness (General disorders) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0 — lethal outcome
Pneumonitis with Septicemia (Infections and infestations) | 0 | 1 — lethal outcome
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — lethal outcome
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — unknown etiology
Neutropenia (Blood and lymphatic system disorders) | 1 | 1
Сervicitis (Reproductive system and breast disorders) | 1 | 0
Hepatic veins compression (Vascular disorders) | 0 | 1
Non-Neutropenic Fever (General disorders) | 0 | 2 — unknown etiology
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchopneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BCD-022 (CJSC BIOCAD) (N=113) | Herceptin ® (F. Hoffmann-La Roche Ltd., Switzerland) (N=110)
Leucopenia (Blood and lymphatic system disorders) | 64 | 54
Leucocytosis (Blood and lymphatic system disorders) | 24 | 35
Neutropenia (Blood and lymphatic system disorders) | 66 | 56
Anemia (Blood and lymphatic system disorders) | 75 | 73
Trombocytopenia (Blood and lymphatic system disorders) | 19 | 21
Elevated absolute neutrophil count (Blood and lymphatic system disorders) | 26 | 29
Elevated hemoglobin (Blood and lymphatic system disorders) | 6 | 11
Lymphopenia (Blood and lymphatic system disorders) | 53 | 40
Lymphocytosis (Blood and lymphatic system disorders) | 14 | 17
Erythropenia (Blood and lymphatic system disorders) | 26 | 25
Erythrocytosis (Blood and lymphatic system disorders) | 12 | 14
Trombocytosis (Blood and lymphatic system disorders) | 27 | 23
Hyperglycemia (Metabolism and nutrition disorders) | 39 | 47
Hyperuricemia (Metabolism and nutrition disorders) | 19 | 24
Elevated alkaline phosphotase (Hepatobiliary disorders) | 28 | 27
Elevated AST (Hepatobiliary disorders) | 29 | 26
Elevated ALT (Hepatobiliary disorders) | 24 | 25
Alopecia (Skin and subcutaneous tissue disorders) | 26 | 26
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 10
Nausea (Gastrointestinal disorders) | 7 | 5
Vomiting (Gastrointestinal disorders) | 6 | 5
Bradypnoea (Respiratory, thoracic and mediastinal disorders) | 15 | 13
Tachypnoea (Reproductive system and breast disorders) | 9 | 8
Neuropathy (Nervous system disorders) | 13 | 9 — non-specified
Elevated urea (Renal and urinary disorders) | 11 | 13
Elevated creatinine (Renal and urinary disorders) | 16 | 14
Arterial hypertension (Vascular disorders) | 13 | 11
Tachycardia (Cardiac disorders) | 22 | 12
Fever (General disorders) | 16 | 14
Generalized weakness (General disorders) | 26 | 25
Elevated lactate degydrohenase (Investigations) | 34 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No